CLINICAL TRIAL: NCT02754284
Title: The Safety and Efficacy Assessment of Functional Collagen Scaffold Transplantation for Larynx Soft Tissue Regeneration
Brief Title: Clinical Study of Regeneration on Larynx Soft Tissue Guided by Functional Collagen Scaffold
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chinese Academy of Sciences (Other Government)
Collaborators: Peking Union Medical College (Other)
Responsible Party: Principal Investigator, Jianwu Dai, Principal Investigator of Regenerative Medicine Laboratory, Institute of Genetics and Developmental Biology, CAS, Chinese Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAS-XDA-LST/IGDB
Record Dates: First submitted 2016-04-19; First posted 2016-04-28 (Estimated); Last update posted 2021-01-05 (Actual); Status verified 2016-04

CONDITIONS: Vocal Cord Dysfunction
MeSH Terms: conditions — Vocal Cord Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Autologous fat transplantation (Experimental)
  Interventions: Biological: Autologous fat transplantation
- Functional collagen scaffold transplantation (Experimental)
  Interventions: Biological: Functional collagen scaffold transplantation

INTERVENTIONS:
Biological: Autologous fat transplantation — Autologous abdominal fat will be injected into vocal cord beneath mucous under surgery microscope.
  Arms: Autologous fat transplantation
Biological: Functional collagen scaffold transplantation — Injectable collagen scaffold combined with adipose derived stem cells that are isolated from abdominal adipose tissue will be injected into vocal cord beneath mucous under surgery microscope.
  Arms: Functional collagen scaffold transplantation

SUMMARY:
This study is carried out to explore the short-term and long-term efficacy of the functional collagen scaffold in guiding laryngeal soft tissue regeneration.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18-65 years old, male or female
2. Severe unilateral vocal cord injury and poor closure of the glottis
3. Disease course was more than 1 year
4. At least two GRBAS scores reach 2 points or more
5. The subjects have read and fully understood the research notes, signed informed consent

Exclusion Criteria:

1. Over speaking professionals, such as teachers, shop assistants.
2. With vital organ dysfunction, such as heart, lung, liver or kidney.
3. Pregnant or lactating women, or in preconception period.
4. Allergic to various drugs.
5. Difficult to be followed-up or cooperate long-termly.
6. Participated in other clinical trials in the last 3 months.
7. With progressive severe disease.
8. Alcoholics or drug addicts.
9. Unable to execute clinical study protocol due to severe mental disorders or lingual barriers
10. With inevitable circumstances of voice damage.
11. Any other unsuitable conditions for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-12; Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Change in subjective auditory perception score | 1 week, 2 week, 1,3,6,12 month after intervention

SECONDARY OUTCOMES:
Change in voice handicap index (VHI) scale | 1 week, 2 week, 1,3,6,12 month after intervention
Objective acoustic evaluation (Jitter) | 1 week, 2 week, 1,3,6,12 month after intervention
Objective acoustic evaluation (Shimmer) | 1 week, 2 week, 1,3,6,12 month after intervention
Objective acoustic evaluation (Normalized noise energy) | 1 week, 2 week, 1,3,6,12 month after intervention
Objective acoustic evaluation（Maximum phonation time） | 1 week, 2 week, 1,3,6,12 month after intervention
Physical status assessment of vocal cords（Motor test of vocal cords） | 1 week, 2 week, 1,3,6,12 month after intervention
Physical status assessment of vocal cords （Closing test of vocal cords） | 1 week, 2 week, 1,3,6,12 month after intervention
Physical status assessment of vocal cords （Morphology of vocal cords） | 1 week, 2 week, 1,3,6,12 month after intervention
Change in volume of vocal cords | 1 week, 2 week, 1,3,6,12 month after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jianwu Dai, Ph.D, Principal Investigator — Chinese Academy of Sciences
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, China